CLINICAL TRIAL: NCT00739011
Title: Validation of Customer Requirements for the HC244/HC254
Brief Title: Validation of HC250 and HC240 Series.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Jessica Hayward, Fisher and Paykel Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FPHC240/250Val
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: SleepStyle 254/244 CPAP series CPAP humidifier

INTERVENTIONS:
Device: SleepStyle 254/244 CPAP series CPAP humidifier — Therapeutic CPAP pressure will be determined for individual subjects during the titration portion of an overnight sleep study. This pressure will range from 4 to 20 cmH20

SUMMARY:
This study is designed to determine the effectiveness of two different CPAP devices. One a standard CPAP which has the ability to store comprehensive compliance and efficacy data and the second a auto adjusting CPAP which uses the energy spectrum analysis of flow signals to automatically adjust CPAP pressure and improve sleep variables.

DETAILED DESCRIPTION:
All patients with suspected obstructive sleep apnea presenting at the Auckland Hospital Sleep Laboratory and referred for either a split-night or full night diagnostic study, will be offered participation in the study and will be recruited. From these patients, a total of 20 patients that are diagnosed with clinical obstructive sleep apnea syndrome, based on diagnostic polysomnography, will undergo titration with the HC254 Auto CPAP. An additional 20 patients will undergo titration with the HC244 CPAP.

The sleep physiologist evaluating the patient clinically will approach patients for participation in this study during their sleep laboratory visit. Consenting patients will undergo either an initial full night diagnostic polysomnography or a split night study as determined by the physician based on clinical requirements. Patients diagnosed with obstructive sleep apnea (AHI > 15/hr) during this diagnostic component will then undergo one of the following:

* Treatment with the HC254 Auto CPAP during the second half of the study.
* Treatment with the HC244 CPAP during the second half of the study.

The sleep physiologist will then determine final CPAP prescriptions for all patients based on the patient's response to CPAP therapy.

5 subjects who have completed the HC254 arm of the study will be brought back to the sleep lab for an additional PSG or partial PSG while on CPAP pressure set to 90th percentile pressure determined on the diagnostic night.

ELIGIBILITY:
Inclusions criteria:

* AHI > 15 on the diagnostic night or portion of the split night study.
* ≥18yrs of age

Exclusion criteria:

* Significant Central Apnea
* CHF
* Co-existing obesity related hypoventilation
* Inability to give informed consent
* Patient intolerance to CPAP
* Anatomical or physiological conditions making CPAP therapy inappropriate.
* Less than 3 hours in the titration period
* Under Land Transport New Zealand (LTNZ) investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | At the end of the sleep study

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Hayward, MSc, Principal Investigator — Fisher and Paykel Healthcare
Locations (2):
- New Zealand (2):
  - Auckland Hospital Sleep laboratory, Auckland
  - Auckland Physiology Sleep Lab, Auckland